CLINICAL TRIAL: NCT00057109
Title: Health Values and Spirituality in Veterans With HIV/AIDS
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: ECI 01-195
Record Dates: First submitted 2003-03-27; First posted 2003-03-28 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2005-12

CONDITIONS: Quality of Life; HIV; Spirituality

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
We have previously shown that: 1) time tradeoff utilities for current health are high, indicating that patients have a strong will to live; 2) half of patients felt that their life was better now than before they were HIV-infected; and 3) certain non-health-related factors such as spirituality and concern and love for one�s children correlated with health values and a sense that life has improved.

DETAILED DESCRIPTION:
Background:

We have previously shown that: 1) time tradeoff utilities for current health are high, indicating that patients have a strong will to live; 2) half of patients felt that their life was better now than before they were HIV-infected; and 3) certain non-health-related factors such as spirituality and concern and love for one�s children correlated with health values and a sense that life has improved.

Objectives:

1) To assess health values of veterans and non-veterans with HIV/AIDS; 2) To characterize spirituality in patients with HIV/AIDS; 3) To derive a power function relating health ratings to utilities; and 4) To assess whether society assigns higher values to health states for veterans than for non-veterans.

Methods:

We interviewed 100 representative veterans with HIV/AIDS from the Cincinnati and Pittsburgh VAMCs and, concurrently, 350 non-veterans with HIV/AIDS from Cincinnati and Washington, DC, twice over 12-18 months. The patient questionnaire included clinical and demographic data; health values measures; a question comparing life now with life before being infected with HIV; and measures of health status/health concerns, HIV symptoms, depressive symptoms, spirituality/religion, adherence, social support, self-esteem, and optimism. We also assessed how medical house officers rate and value the health state of a hypothetical patient with congestive heart failure, identified either as a 72-year-old veteran or merely as a 72-year-old male.

Status:

Data collection completed ahead of schedule. Several manuscripts published with others to be submitted soon.

ELIGIBILITY:
Inclusion Criteria:

Adults with HIV/AIDS

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Tsevat, MD MPH, Principal Investigator — Cincinnati VA Medical Center, Cincinnati, OH
Locations (2):
- United States (2):
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Sherman SN, Mrus JM, Yi MS, Feinberg J, Tsevat J. How do patients with HIV/AIDS understand and respond to health value questions? J Gen Intern Med. 2006 Dec;21 Suppl 5(Suppl 5):S56-61. doi: 10.1111/j.1525-1497.2006.00647.x. PMID 17083502
- [Result] Cotton S, Puchalski CM, Sherman SN, Mrus JM, Peterman AH, Feinberg J, Pargament KI, Justice AC, Leonard AC, Tsevat J. Spirituality and religion in patients with HIV/AIDS. J Gen Intern Med. 2006 Dec;21 Suppl 5(Suppl 5):S5-13. doi: 10.1111/j.1525-1497.2006.00642.x. PMID 17083501
- [Result] Kudel I, Farber SL, Mrus JM, Leonard AC, Sherman SN, Tsevat J. Patterns of responses on health-related quality of life questionnaires among patients with HIV/AIDS. J Gen Intern Med. 2006 Dec;21 Suppl 5(Suppl 5):S48-55. doi: 10.1111/j.1525-1497.2006.00645.x. PMID 17083500
- [Result] Cotton S, Tsevat J, Szaflarski M, Kudel I, Sherman SN, Feinberg J, Leonard AC, Holmes WC. Changes in religiousness and spirituality attributed to HIV/AIDS: are there sex and race differences? J Gen Intern Med. 2006 Dec;21 Suppl 5(Suppl 5):S14-20. doi: 10.1111/j.1525-1497.2006.00641.x. PMID 17083495
- [Result] Mrus JM, Leonard AC, Yi MS, Sherman SN, Fultz SL, Justice AC, Tsevat J. Health-related quality of life in veterans and nonveterans with HIV/AIDS. J Gen Intern Med. 2006 Dec;21 Suppl 5(Suppl 5):S39-47. doi: 10.1111/j.1525-1497.2006.00644.x. PMID 17083499
- [Result] Tsevat J, Leonard AC, Szaflarski M, Sherman SN, Cotton S, Mrus JM, Feinberg J. Change in quality of life after being diagnosed with HIV: a multicenter longitudinal study. AIDS Patient Care STDS. 2009 Nov;23(11):931-7. doi: 10.1089/apc.2009.0026. PMID 19821724
- [Result] Szaflarski M, Ritchey PN, Leonard AC, Mrus JM, Peterman AH, Ellison CG, McCullough ME, Tsevat J. Modeling the effects of spirituality/religion on patients' perceptions of living with HIV/AIDS. J Gen Intern Med. 2006 Dec;21 Suppl 5(Suppl 5):S28-38. doi: 10.1111/j.1525-1497.2006.00646.x. PMID 17083497
- [Result] Yi MS, Mrus JM, Wade TJ, Ho ML, Hornung RW, Cotton S, Peterman AH, Puchalski CM, Tsevat J. Religion, spirituality, and depressive symptoms in patients with HIV/AIDS. J Gen Intern Med. 2006 Dec;21 Suppl 5(Suppl 5):S21-7. doi: 10.1111/j.1525-1497.2006.00643.x. PMID 17083496